CLINICAL TRIAL: NCT03868488
Title: Mental Imagery Tasks to Reduce IGD Cravings: Visual Imagery and Auditory Imagery
Brief Title: Mental Imagery Tasks to Reduce Internet Gaming Disorder (IGD) Cravings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jin-tao Zhang (Other)
Responsible Party: Sponsor-Investigator, Jin-tao Zhang, Associated Professor, Beijing Normal University
Organization: Beijing Normal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Mental imagery tasks
Record Dates: First submitted 2019-03-01; First posted 2019-03-11 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Internet Gaming Disorder
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual imagery tasks group (Experimental): During the intervention, each participant of this group will be asked to create visual mental images.
  Interventions: Behavioral: Imagery tasks
- Auditory imagery tasks group (Experimental): During the intervention, each participant of this group will be asked to create auditory mental images.
  Interventions: Behavioral: Imagery tasks

INTERVENTIONS:
Behavioral: Imagery tasks — All participants need to finish both visual imagery tasks and auditory imagery tasks. Visual imagery tasks and auditory imagery tasks will be carried out at intervals to avoid the influence of different tasks. The sequence of imagery tasks will be counterbalanced across participants.

SUMMARY:
To test whether visual and auditory imagery tasks can effectively reduce the craving for IGD.

DETAILED DESCRIPTION:
This project is to use imagery tasks to reduce the craving of internet gamers. To test whether visual and auditory imagery tasks can effectively reduce the craving for IGD. This project will be conducted in Beijing, China, based on a large sample of internet gamers.

ELIGIBILITY:
Inclusion Criteria:

* The scores of the 9 items of The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition(DSM-5) recommended diagnosis for Internet gaming disorder ≥ 5.
* Engagement in popular Internet games (e.g. Arena of Valor, League of Legends and Player Unknown's Battle Grounds) for over 20 hours per week for a minimum of 12 months.
* The scores of the Young-Internet Addiction Test(Y-IAT) ≥ 50

Exclusion Criteria:

* Current or history of use of illegal substances and gambling;
* Current or history of psychiatric or neurological illness;
* Current use of psychotropic medications.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-10 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
The craving of internet gamers | 0-1 minutes before each set of cue
  The craving of internet gamers is measured by a single item Visual Analogue Scale with 1 to 7 likert score
The craving of internet gamers after cue | 0-1 minutes after showing cue
  The craving of internet gamers is measured by a single item Visual Analogue Scale with 1 to 7 likert scoreScale with 1 to 7 likert score
The craving of internet gamers | 0-1 minutes after finishing each block of tasks
  The craving of internet gamers is measured by a single item Visual Analogue Scale with 1 to 7 likert score

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tao Zhang, PhD, Principal Investigator — Beijing Normal University
Locations (1):
- State Key Laboratory of Cognitive Neuroscience and Learning, Beijing Normal University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] May J, Andrade J, Panabokke N, Kavanagh D. Visuospatial tasks suppress craving for cigarettes. Behav Res Ther. 2010 Jun;48(6):476-85. doi: 10.1016/j.brat.2010.02.001. Epub 2010 Feb 7. PMID 20189549
- [Background] Yates M, Kamboj SK. Alcohol related mental imagery: The effects of a priming dose in at risk drinkers. Addict Behav Rep. 2017 Aug 31;6:71-75. doi: 10.1016/j.abrep.2017.08.003. eCollection 2017 Dec. PMID 29450239